CLINICAL TRIAL: NCT04162340
Title: CD4-specific CAR T Cells (CD4 CAR T Cells) for Relapsed/Refractory T Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: iCAR Bio Therapeutics Ltd. (Industry); Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICG155-001
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: T Cell Lymphoma in Relapse; Refractory T-Cell Lymphoma
Keywords: CD4-specific CAR T; T cell leukemia; T cell lymphoma; CD4CAR
MeSH Terms: conditions — Lymphoma, T-Cell; Leukemia, T-Cell

STUDY DESIGN:
Intervention Model Description: Dose escalation phase: CD4 CAR T cells transduced with a lentiviral vector to express CD4 chimeric receptor domain on T cells with an escalation approach, 2e6 to 5e6 CAR-T cells/kg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD4 CAR T cells (Experimental): Dose escalation phase: CD4 CAR T cells transduced with a lentiviral vector to express CD4 chimeric receptor domain on T cells with an escalation approach, 2e6 to 5e6 CAR-T cells/kg
  Interventions: Biological: CD4 CAR T cells

INTERVENTIONS:
Biological: CD4 CAR T cells — CD4 CAR T cells administered to patients, will be either fresh or thawed CAR T cells by IV injection after receiving lymphodepleting chemotherapy.

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of CD4 CAR T cells in patients with relapsed and/or refractory T cell lymphoma.

DETAILED DESCRIPTION:
CD4-specific CAR is a chimeric antigen receptor immunotherapy treatment designed to treat lymphoma/leukemia expressing CD4 antigen. CD4+ T cell lymphomas are a subset of leukemias and lymphomas that are positive for the surface protein CD4. The purpose of this study is to evaluate the efficacy and safety of CD4 CAR T cells.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent; Patients volunteer to participate in the research
* Diagnosis is mainly based on the World Health Organization (WHO) 2008
* Patients have exhausted standard therapeutic options
* Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 1 weeks
* Female must be not pregnant during the study

Exclusion Criteria:

* Patients declining to consent for treatment
* Prior solid organ transplantation
* Potentially curative therapy including chemotherapy or hematopoietic cell transplant
* Any drug used for GVHD must be stopped >1 week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events after CD4 CAR T cells cell infusion | 2 years particularly the first 28 days after infusion
  Determine the toxicity profile of CD4 CAR T cell therapy

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | up to 6 months
  Incidence of treatment-emergent adverse events
Disease Free Survival (DFS) | up to 2 years
  Disease Free Survival (DFS) (IMWG criteria)
Progression-Free Survival (PFS) | up to 2 years
  Progression-Free Survival (IMWG criteria)
Overall Survival (OS) | up to 2 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Zhang, MD/PhD, Principal Investigator — Peking University Shenzhen Hospital, China; Fang Liu, MD/PhD, Principal Investigator — Chengdu Military Hospital
Locations (2):
- China (2):
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Chengdu Military General Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No